CLINICAL TRIAL: NCT04763980
Title: Navigate Study: Use of a Community-Based Health Coach to Improve Access to Germline Genetic Testing Among African American Men With Prostate Cancer
Brief Title: Community-Based Health Coach for Access to Germline Genetic Testing Among African American Men With Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Lazarex Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 20553; NCI-2021-01027 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Genetic Testing; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CLOSED TO ENROLLMENT - Initial Pilot Cohort A (survey, genetic testing) (Active Comparator): Participants complete a survey about knowledge of, attitudes towards, and awareness of genetic testing and technology preferences and use over 30 minutes at baseline and over 20 minutes at exit or follow up. Participants may also undergo genetic testing.
  Interventions: Other: Genetic Testing; Other: Survey Administration
- CLOSED TO ENROLLMENT -Initial Pilot Cohort B (educational session, survey, genetic testing) (Experimental): Participants engage in educational session with health coach over 60 minutes. Participants also complete a survey about knowledge of, attitudes towards, and awareness of genetic testing and technology preferences and use over 30 minutes at baseline and over 20 minutes at exit or follow up. Participants may undergo genetic testing. Participant and provider interviews will be conducted at end of study.
  Interventions: Other: Educational Intervention; Other: Genetic Testing; Other: Survey Administration
- Part 1 (educational session, survey, genetic testing) (Experimental): Participants engage in educational session lasting 15-30 minutes with health coach in-person or remotely who will be using a ProGene chatbot to augment the session over 15-30 minutes. Participants also complete surveys about knowledge of, attitudes towards, and awareness of genetic testing and technology preferences. Participants may undergo genetic testing.
  Interventions: Other: Educational Intervention; Other: Genetic Testing; Other: Survey Administration; Other: ProGene Artificial Intelligence (AI) Platform; Other: Interviews
- Part 2 Pilot (educational session, survey, genetic testing) (Experimental): Clinical participants engage in educational session lasting about 15-30 minutes with health coach in-person or remotely who will be using a ProGene chatbot to augment the session. Participants also complete surveys about knowledge of, attitudes towards, and awareness of genetic testing and technology preferences. Community and clinical participants may undergo genetic testing.
  Interventions: Other: Educational Intervention; Other: Genetic Testing; Other: Survey Administration; Other: ProGene Artificial Intelligence (AI) Platform; Other: Interviews

INTERVENTIONS:
Other: Educational Intervention — Participate in educational session with health coach
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: CLOSED TO ENROLLMENT -Initial Pilot Cohort B (educational session, survey, genetic testing); Part 1 (educational session, survey, genetic testing); Part 2 Pilot (educational session, survey, genetic testing)
Other: Genetic Testing — Undergo genetic testing
  Other Names: Genetic analysis; Genetic Examination; Genetic Test
Other: Survey Administration — Complete surveys throughout course of study.
  Other Names: Questionnaire Administration
Other: ProGene Artificial Intelligence (AI) Platform — AI Platform to be used by health coach during sessions
  Other Names: ProGene AI Platform; ProGene
  Arms: Part 1 (educational session, survey, genetic testing); Part 2 Pilot (educational session, survey, genetic testing)
Other: Interviews — Participant and provider interviews will be conducted by study staff.
  Other Names: Participant interviews
  Arms: Part 1 (educational session, survey, genetic testing); Part 2 Pilot (educational session, survey, genetic testing)

SUMMARY:
This clinical trial studies barriers to genetic testing in African American men with prostate cancer and whether tailored, culturally relevant genetic testing education provided by a community-based health coach is beneficial in improving knowledge, attitudes, and awareness of genetic testing. Information gained from this study, may help researchers better understand and learn more about how to increase access to germline genetic testing in underrepresented populations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess uptake of genetic testing using tailored education strategies and culturally relevant cancer resources delivered by a community-based health coach (Initial Pilot Cohorts).

II. To assess barriers to the intervention (Part 1). III. To evaluate consent rate of germline testing among participants receiving the intervention (Part 2).

SECONDARY OBJECTIVES:

I. To assess decisional conflict among African American men receiving tailored education strategies and culturally relevant cancer resources on genetic testing delivered by a community-based health coach (Initial Pilot Cohorts).

II. To assess facilitators to the intervention (Part 1).

III. To assess acceptability of the intervention (Parts 1 and 2).

IV. To characterize patient and health coach use of ProGene (Part 1).

V. To evaluate completion rate of germline testing among participants receiving the intervention (Part 2).

VI. To evaluate change in participant knowledge about germline testing among patient participants (Part 2).

VII. To evaluate change in participant attitudes toward germline testing among patient participants (Part 2).

VIII. To evaluate change in decisional conflict about germline testing among patient participants (Part 2).

IX. To evaluate reach of the intervention (Part 2).

X. To evaluate barriers and facilitators to the intervention (Part 2).

XI. To identify reasons for declining germline testing.

TERTIARY OBJECTIVE:

I. To assess the germline mutation rate among African American men with prostate cancer (Initial Pilot Cohorts)

OUTLINE: The initial pilot phase of the study has concluded. Participants are assigned to Parts 1 or 2 of current study.

CLOSED TO ENROLLMENT: INITIAL PILOT COHORT A:

Participants complete a survey about knowledge of, attitudes towards, and awareness of genetic testing and technology preferences and use over 30 minutes at baseline and over 20 minutes at exit or follow up. Participants may also undergo genetic testing.

CLOSED TO ENROLLMENT: INITIAL PILOT COHORT B:

Participants engage in an educational session with health coach over 60 minutes. Participants also complete a survey about knowledge of, attitudes towards, and awareness of genetic testing and technology preferences and use over 30 minutes at baseline and over 20 minutes at exit or follow up. Participants may undergo genetic testing.

PART 1:

Participants engage in an educational session with health coach over 60 minutes. Participants also complete a survey about knowledge of, attitudes towards, and awareness of genetic testing and technology preferences and use over 30 minutes at baseline and over 20 minutes at exit or follow up. Participants may undergo genetic testing.

PART 2:

Participants in this secondary pilot engage in an educational session with health coach over 60 minutes. Participants also complete a survey about knowledge of, attitudes towards, and awareness of genetic testing and technology preferences and use over 30 minutes at baseline and over 20 minutes at exit or follow up. Participants may undergo genetic testing.

ELIGIBILITY:
Inclusion Criteria:

CLOSED TO ENROLLMENT: INITIAL PILOT COHORT:

Participants:

1. Age >=18 years old.
2. Able to speak and read in English.
3. Have no known cancer risk genetic mutation.
4. Self-identify as Black or African American.
5. Self-report a diagnosis of regional (lymph node positive), advanced, or metastatic prostate cancer per National Comprehensive Cancer Network (NCCN) guidelines.

ENROLLING: PART 1:

Participants:

1. Age >=18 years old.
2. Able to speak and read in English.
3. Able to understand study procedures and to comply with them for the entire length of the study.
4. Able to verbally consent.
5. Self-identifies as Black or African-American.
6. Self-reports a diagnosis of regional (lymph node positive), advanced, or metastatic prostate cancer.

Note: Participants may or may not have had germline testing in the past, as a range of experiences is valuable for holistic feedback.

Providers:

1. Self-identifies as a medical oncologist or genetics provider.
2. Able to speak and read in English.
3. Able to understand study procedures and to comply with them for the entire length of the study.
4. Able to verbally consent.

ENROLLING: PART 2:

Participants:

1. Age >=18 years old.
2. Able to speak and read in English.
3. Able to understand study procedures and to comply with them for the entire length of the study.
4. Able to provide written informed consent.
5. Have no known cancer risk genetic mutation.
6. Self-identify as Black or African American.
7. Self-report a diagnosis of regional (lymph node positive), advanced, or metastatic prostate cancer per NCCN guidelines.
8. For patients recruited from the clinic: Presence of an oncology appointment within 3 months where germline testing will be discussed.

Exclusion Criteria:

CLOSED TO ENROLLMENT: INITIAL PILOT COHORT.

1. Prior germline genetic test.
2. Age <18 years old.
3. Unable to read or answer forms.

ENROLLING: PART 1:

1. Contraindication to any study-related procedure or assessment.

ENROLLING: PART 2:

1. Self-reports prior germline genetic test.
2. Contraindication to any study-related procedure or assessment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Consent rate for germline testing (Initial Pilot Cohort and Part 2) | At baseline (1 day)
  The consent rate for each cohort will be defined as proportion of patients enrolled in the study who agree to undergo germline genetic testing with Color genomics. The point estimate and 90% confidence interval will be provided.
Frequency of reported barriers to interventions (Part 1) | Up to 30 days
  Participant- and provider-reported barriers to engaging in the intervention for participants to make an informed decision about germline testing will be reported descriptively.

SECONDARY OUTCOMES:
Decisional conflict scale score (Initial Pilot Cohort and Part 2) | Up to 120 days
  The decisional conflict scale will be scored using a validated instrument. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict). Summary statistics with median and interquartile range will be obtained.
Frequency of reported facilitators to interventions (Part 1 and 2) | Up to 120 days
  Participant- and provider-reported facilitators to engaging in the intervention for participants to make an informed decision about germline testing.
Mean score of theoretical framework of acceptability (TFA) questionnaire (Part 1 and Part 2) | Up to 120 days
  Participant-reported acceptability of the intervention will be described using the TFA questionnaire. Scores on the TFA items will be averaged across all participants. Items will be scored on a 5-point scale: 1= Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5= Completely agree. All negatively worded items will be reverse-scored for a total score of 24-120. Higher scores represent greater acceptability (more positive attitudes). The mean score and standard deviation will be reported.
Number of recorded inputs into ProGene (Part 1) | Up to 30 days
  The number of recorded data inputs into the ProGene platform will be reported descriptively to characterize patient-participant and health coach use of ProGene.
Proportion of patient participants who complete germline testing (Part 2) | Up to 120 days
  The completion rate is defined as the proportion of patient-participants who complete germline testing within 90 days of intervention will be reported.
Mean score of adapted KnowGene germline testing knowledge survey (Part 2) | Up to 120 days
  Knowledge of tumor genetic testing adapted from a validated survey from Blanchette, et al.+ select questions from a survey from Rogith, et al. will be utilized to measure the level of cancer genomic testing knowledge. "Don't know" will be scored as incorrect. The proportion of correct responses will be calculated to generate a total score between 0-100, with a higher score indicating greater knowledge. No items will be weighted. Since all items are required, we anticipate missing responses will be rare. Any missing data will be managed case-by-case post-hoc.
Mean score of genetic testing attitudes survey (Part 2) | Up to 120 days
  Attitude and expectations measure for tumor genetic testing is a 17-item measure adapted from a validated survey from Blanchette, et al. including one open-ended investigator-created item. Items on the attitude scoring scale range from "Yes" = 1 and "No" or "Unsure" = 0
Proportion of individuals classified as "supporters" (Part 2) | Up to 120 days
  Proportion of individuals classified as "supporters" of genetic testing
Proportion of participants who consent to study (Part 2) | Up to 120 days
  Proportion of participants who consent to study among those approached as potential participants will be reported
Frequency of reported barriers to interventions (Part 2) | Up to 120 days
  Participant- and provider-reported barriers to engaging in the intervention for participants to make an informed decision about germline testing will be reported descriptively.
Frequency of reasons for declining testing (Part 2) | Up to 120 days
  Patient-participant reported reasons for declining germline testing will be reported descriptively.

OTHER OUTCOMES:
Highly penetrant germline genetic mutation rate and variants of unknown significance among all participants who undergo germline testing | At baseline and exit/follow-up visit (up to 2 days)
  Will be determined by the sum of all alterations detected on Color genomics. Summary statistics will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kwon, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - San Francisco Veterans Administration Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No